CLINICAL TRIAL: NCT02198547
Title: Evaluation of Magnesium as Adjuvant to Ropivacaine for Sciatic Block at Popliteal Level.
Brief Title: Magnesium as Adjuvant for Sciatic Block
Acronym: Mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, MD, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CarGalMg
Record Dates: First submitted 2014-03-17; First posted 2014-07-23 (Estimated); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Hallux Valgus
Keywords: Local anesthetic adjuvant,; Magnesium solfatus,; Sciatic block
MeSH Terms: conditions — Hallux Valgus | interventions — Magnesium Sulfate; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine Magnesium sulfate (Experimental): Locoregional anesthesia for valgus allux correction with ropivacaine 7,5 mg/ml and Mg 4 mg/Kg.
  Sciatic block at popliteal level.
  Interventions: Drug: Magnesium Sulfate
- Ropivacaine (Active Comparator): Patients undergoing allux valgus correction with locoregional anesthesia with ropivacaine 7,5 mg/ml, without MG
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate — Mg used with ropivacaine for sciatic nerve blick
  Arms: Ropivacaine Magnesium sulfate
Drug: Ropivacaine — Ropivacaine 7,5 mg/ml used for sciatic nerve block
  Arms: Ropivacaine

SUMMARY:
The aim of the study is to evaluate if Magnesium added to ropivacaine can reduce onset time and can enhance offset time.

DETAILED DESCRIPTION:
Patients are randomly divided into two groups: group "M" (Ropivacaina 7,5 mg/ml with Mg 4 mg/Kg)and group"C" (without Mg).

Standard monitoring is applied to each patient in perioperative period. An indipendent observer collect data: time to perform block, sensitivity onset,motor onset, pain during surgery and complication.

In the post-operative period till 24 hours for each patient is evaluated off-set time, pain and analgesic consumption.

ELIGIBILITY:
Inclusion Criteria:

* given consent
* allux valgus correction surgery

Exclusion Criteria:

* allergy to local anesthetic
* infection in the site of puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Mg as adjuvant to local anesthetic | Till 24 hours
  We evaluate if Mg affects onset and offset time of ropivacaine 7,5 mg/ml in sciatic block at popliteal level

SECONDARY OUTCOMES:
Post-operative pain | 3 hours
  We evaluate post-operative pain at rest and in movement at 3-6-12-24 hours with NRS scale
Post-operative analgesic consumption | till 24 hours
  We evaluate consumption of opioid and non-opioid analgesic used in the post-operative period.
Post-operative pain | 6 hours
  Evaluation of pain with NRS scale
post-operative pain | 12 hours
  Evaluation of pain with NRS scale
Post-operative pain | 24 hours
  Evaluation of pain with NRS scale

OTHER OUTCOMES:
Patients' approval | At 24 hours
  We evaluate the grade of approval of patients with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, MD, Principal Investigator — Campus Bio Medico
Locations (1):
- Campus Bio-Medico, Rome, Italy

REFERENCES:
- [Background] Lee AR, Yi HW, Chung IS, Ko JS, Ahn HJ, Gwak MS, Choi DH, Choi SJ. Magnesium added to bupivacaine prolongs the duration of analgesia after interscalene nerve block. Can J Anaesth. 2012 Jan;59(1):21-7. doi: 10.1007/s12630-011-9604-5. Epub 2011 Oct 20. PMID 22012543
- [Background] Ekmekci P, Bengisun ZK, Akan B, Kazbek BK, Ozkan KS, Suer AH. The effect of magnesium added to levobupivacaine for femoral nerve block on postoperative analgesia in patients undergoing ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2013 May;21(5):1119-24. doi: 10.1007/s00167-012-2093-4. Epub 2012 Jun 14. PMID 22696144
- [Background] Dogru K, Yildirim D, Ulgey A, Aksu R, Bicer C, Boyaci A. Adding magnesium to levobupivacaine for axillary brachial plexus block in arteriovenous fistule surgery. Bratisl Lek Listy. 2012;113(10):607-9. doi: 10.4149/bll_2012_136. PMID 23094900
- [Background] Vastani N, Seifert B, Spahn DR, Maurer K. Sensitivities of rat primary sensory afferent nerves to magnesium: implications for differential nerve blocks. Eur J Anaesthesiol. 2013 Jan;30(1):21-8. doi: 10.1097/EJA.0b013e32835949ab. PMID 23138572
- [Background] Bailard NS, Ortiz J, Flores RA. Additives to local anesthetics for peripheral nerve blocks: Evidence, limitations, and recommendations. Am J Health Syst Pharm. 2014 Mar 1;71(5):373-85. doi: 10.2146/ajhp130336. PMID 24534592